CLINICAL TRIAL: NCT05032872
Title: Social Exergame Intervention to Promote Physical Activity, Social Support, And Well-Being in Family Caregivers
Brief Title: Exergame Study for Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GoGrowExergrame #20104R; P30AG048785 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-10

CONDITIONS: Sedentary Lifestyle
Keywords: Family Caregivers
MeSH Terms: conditions — Sedentary Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Exergame Treatment Group (Experimental): The treatment group will wear a Fitbit step counter for 8 weeks. In addition, participants will use the full version of the Go&Grow fitness app for 6 weeks.
  Interventions: Behavioral: Social Exergame Treatment Group
- Control Group (Active Comparator): The control group will wear a Fitbit step counter for 8 weeks. In addition, participants will use the Go&Grow fitness app without the social features for 6 weeks.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Social Exergame Treatment Group — * Physical activity tracking, walk to grow flowers and plant their own garden
  * Follow workout tutorials
  * Daily steps tracked by Fitbit and workout log tracked by the app
  * Daily reminders to wear Fitbit, use the app, and share stories to unlock new flowers to grow
  * Includes social features: like, reply, and see other's stories, and share their stories; Access to other people's gardens
  * In-app rewards (unlock new flowers to grow each week) if participants post stories
  Arms: Social Exergame Treatment Group
Behavioral: Control Group — * Physical activity tracking, walk to grow flowers and plant their own garden
  * Follow workout tutorials
  * Daily steps tracked by Fitbit and workout log tracked by the app
  * Daily reminders to wear Fitbit and use the app
  Arms: Control Group

SUMMARY:
The goal of this study is to examine Go&Grow as a social exergame intervention to increase physical activity and social support, to promote well-being in family caregivers, and to test social support and physical activity as mechanisms for the effects of the intervention.

DETAILED DESCRIPTION:
The study is a 2-week baseline and 6-week intervention aimed at comparing the feasibility and efficacy of an exergame (Go&Grow without social contact components) and a social exergame (full version of Go&Grow) in promoting physical activity, social support, and well-being in family caregivers. The study also seeks to test social support and physical activity as mechanisms for the relationships between condition (exergame non-social vs social exergame) and wellbeing. Participants will be randomly assigned using a random assignment generator to either the control condition (exergame non-social) or the treatment condition (social exergame) on a rolling basis. Participants from both conditions will be reminded daily via app-based notifications during the intervention period to wear their Fitbit and to play the game.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are caregivers for a family member (e.g., relative, spouse, friend) who is 65 years or older and is either frail, has a disability, or has at least one chronic illness
* 40 years or older
* Own an Android smartphone with Google play store/internet access
* Able to walk for at least 20 minutes at a time
* Comfortable wearing a fitness tracker for the duration of the study
* Familiar with smartphone app usages
* Comfortable with using the study-related app for the duration of the study

Exclusion Criteria:

* Had a recent (within the past 6 months) cardiovascular event or fall.
* Currently participating in any other physical activity study/intervention
* Currently own or use a Fitbit or other activity tracking watches
* Knows someone who is participating or has participated in the study
* Currently physically active (exercise regularly 3 times a week or more for at least 30 minutes)
* More than 2 errors on the Short Portable Mental Status Questionnaire (Pfeiffer, 1975).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brandeis University, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin XY, Zhang L, Yoon S, Zhang R, Lachman ME. A Social Exergame Intervention to Promote Physical Activity, Social Support, and Well-Being in Family Caregivers. Gerontologist. 2023 Oct 17;63(9):1456-1466. doi: 10.1093/geront/gnad028. PMID 36916022

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 80 participants enrolled (agreed to participate in the study following completion of informed consent), and were all assigned to each arm/group. However, only 38/42 people assigned in the control group completed the pretest, thus we don't have complete pretest data for 4 people in the control group, and 2 of these 4 people didn't complete any demographic information, so we don't have their baseline characteristic measures.
Groups:
- Social Exergame Treatment Group: The treatment group will wear a Fitbit step counter for 8 weeks. In addition, participants will use the full version of the Go&Grow fitness app for 6 weeks.
  Social Exergame Treatment Group: - Physical activity tracking, walk to grow flowers and plant their own garden
  * Follow workout tutorials
  * Daily steps tracked by Fitbit and workout log tracked by the app
  * Daily reminders to wear Fitbit, use the app, and share stories to unlock new flowers to grow
  * Includes social features: like, reply, and see other's stories, and share their stories; Access to other people's gardens
  * In-app rewards (unlock new flowers to grow each week) if participants post stories
- Control Group: The control group will wear a Fitbit step counter for 8 weeks. In addition, participants will use the Go&Grow fitness app without the social features for 6 weeks.
  Control Group: - Physical activity tracking, walk to grow flowers and plant their own garden
  * Follow workout tutorials
  * Daily steps tracked by Fitbit and workout log tracked by the app
  * Daily reminders to wear Fitbit and use the app
Period: Overall Study
Arm/Group | Social Exergame Treatment Group | Control Group
Started (enrolled in the study) | 38 | 42
Completed Pretest | 38 | 38
Completed (completed posttest) | 31 | 35
Not Completed | 7 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: Not all participants answered all questions/questionnaires because they were allowed to skip questions hence the discrepancy of sample size between measures.
  Many of the weekly measures had missing data as not all participants completed the weekly survey or had weekly steps. 2 out of the 40 completed demographic but dropped out before taking the pretest.
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Exergame Treatment Group | Control Group | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.71 (10.04) | 57.03 (11.99) | 56.38 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 65
  Male | 3 | 10 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 36 | 36 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 24 | 33 | 57
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Steps
Description: Steps were automatically synced from the Fitbit for both conditions daily. Days with 500 or fewer recorded steps were coded as missing. Weekly step averages were calculated for weeks with 4 or more days not coded missing. The first two weeks of baseline steps were averaged to form the baseline step.
  Percent change of steps was calculated as the difference between the average weekly steps during the intervention (weeks 3-8) and baseline steps divided by baseline steps.
Time Frame: Percent Change of Steps from baseline to Weeks 3, 4, 5, 6, 7, and 8
Population: some weeks were coded as missing since not all participants recorded steps for all weeks
Measure: Mean (Standard Deviation); unit: Percent Change of Steps from Baseline
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 31 | 33
Percent Change of Steps from Baseline
  Percent Change From Baseline to Week 3 | 4.68 (29) | 4.77 (23)
  Percent Change From Baseline to Week 4: number analyzed (Participants) | 30 | 33
  Percent Change From Baseline to Week 4 | 11.87 (33) | 2.69 (22)
  Percent Change From Baseline to Week 5: number analyzed (Participants) | 30 | 33
  Percent Change From Baseline to Week 5 | 10 (46) | 11.11 (26)
  Percent Change From Baseline to Week 6: number analyzed (Participants) | 29 | 33
  Percent Change From Baseline to Week 6 | 5.33 (38) | 11.26 (28)
  Percent Change From Baseline to Week 7: number analyzed (Participants) | 30 | 33
  Percent Change From Baseline to Week 7 | 3.11 (35) | 5.66 (33)
  Percent Change From Baseline to Week 8: number analyzed (Participants) | 27 | 30
  Percent Change From Baseline to Week 8 | 10 (48) | -6.45 (24)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time by condition interaction; Test type: Superiority; p = .49, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

2. Primary Outcome: Lubben Social Network Scale (LSNS)
Description: Self-report measure of social support from the Lubben Social Network Scale for family and friends with scores summed across 18 items. Possible scores range from 0-60, with higher scores indicating higher social support.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Pretest | 32.32 (7.98) | 30.64 (9.26)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 32.23 (9.81) | 28.40 (9.15)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .48, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

3. Primary Outcome: Social Connectedness Scale
Description: Social Connectedness Scale was administered weekly during the intervention with the following subscales:
  relationship salience, shared understandings, knowing other's experiences, satisfaction with the contact quantity and quality, and dissatisfaction with contact quantity. Scores were averaged across items from each subscale and possible scores ranged from 1 to 7 with higher scores indicating a higher level of the subscale.
Time Frame: Baseline (Average of Week 1 and 2), Weekly during the intervention from Week 3 to 8
Population: not all participants completed each weekly survey. There were missing weekly surveys for some participants on some weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Knowing Others' Experience Baseline (Average of Week 1 and 2) | 4.88 (.92) | 4.72 (1.06)
  Knowing Others' Experience Week 3: number analyzed (Participants) | 33 | 36
  Knowing Others' Experience Week 3 | 4.7 (1.22) | 4.72 (1.18)
  Knowing Others' Experience Week 4: number analyzed (Participants) | 30 | 36
  Knowing Others' Experience Week 4 | 4.96 (1.23) | 4.87 (1.12)
  Knowing Others' Experience Week 5: number analyzed (Participants) | 31 | 35
  Knowing Others' Experience Week 5 | 4.85 (1.4) | 4.67 (1.17)
  Knowing Others' Experience Week 6: number analyzed (Participants) | 32 | 35
  Knowing Others' Experience Week 6 | 5 (1.14) | 4.67 (1.28)
  Knowing Others' Experience Week 7: number analyzed (Participants) | 29 | 34
  Knowing Others' Experience Week 7 | 4.63 (1.22) | 4.66 (1.27)
  Knowing Others' Experience Week 8: number analyzed (Participants) | 32 | 35
  Knowing Others' Experience Week 8 | 4.77 (1.31) | 4.70 (1.33)
  Relationship Salience Baseline (Average of Week 1 and 2) | 4.55 (1.22) | 4.47 (1.36)
  Relationship Salience Week 3: number analyzed (Participants) | 33 | 36
  Relationship Salience Week 3 | 4.60 (1.37) | 4.46 (1.33)
  Relationship Salience Week 4: number analyzed (Participants) | 30 | 36
  Relationship Salience Week 4 | 4.82 (1.19) | 4.59 (1.21)
  Relationship Salience Week 5: number analyzed (Participants) | 31 | 35
  Relationship Salience Week 5 | 4.69 (1.21) | 4.71 (1.32)
  Relationship Salience Week 6: number analyzed (Participants) | 32 | 35
  Relationship Salience Week 6 | 4.80 (1.34) | 4.64 (1.36)
  Relationship Salience Week 7: number analyzed (Participants) | 29 | 34
  Relationship Salience Week 7 | 4.79 (1.23) | 4.74 (1.24)
  Relationship Salience Week 8: number analyzed (Participants) | 32 | 35
  Relationship Salience Week 8 | 4.79 (1.14) | 4.57 (1.28)
  Satisfaction with contact quality Baseline (Average of Week 1 and 2) | 4.71 (1.44) | 4.69 (1.63)
  Satisfaction with contact quality week 3: number analyzed (Participants) | 33 | 36
  Satisfaction with contact quality week 3 | 4.98 (1.55) | 4.69 (1.85)
  Satisfaction with contact quality week 4: number analyzed (Participants) | 30 | 36
  Satisfaction with contact quality week 4 | 4.96 (1.45) | 4.66 (1.76)
  Satisfaction with contact quality week 5: number analyzed (Participants) | 31 | 35
  Satisfaction with contact quality week 5 | 5.01 (1.6) | 4.77 (1.79)
  Satisfaction with contact quality week 6: number analyzed (Participants) | 32 | 35
  Satisfaction with contact quality week 6 | 5.18 (1.46) | 4.84 (1.76)
  Satisfaction with contact quality week 7: number analyzed (Participants) | 29 | 34
  Satisfaction with contact quality week 7 | 5.23 (1.48) | 4.72 (1.90)
  Satisfaction with contact quality week 8: number analyzed (Participants) | 32 | 35
  Satisfaction with contact quality week 8 | 5.21 (1.44) | 4.57 (1.95)
  Dissatisfaction with contact quantity Baseline (Average of Week 1 and 2) | 3.98 (1.29) | 4.47 (1.42)
  Dissatisfaction with contact quantity week 3: number analyzed (Participants) | 33 | 36
  Dissatisfaction with contact quantity week 3 | 4.16 (1.49) | 4.41 (1.52)
  Dissatisfaction with contact quantity week 4: number analyzed (Participants) | 30 | 36
  Dissatisfaction with contact quantity week 4 | 3.88 (1.45) | 4.34 (1.59)
  Dissatisfaction with contact quantity week 5: number analyzed (Participants) | 31 | 35
  Dissatisfaction with contact quantity week 5 | 3.78 (1.40) | 4.37 (1.63)
  Dissatisfaction with contact quantity week 6: number analyzed (Participants) | 32 | 35
  Dissatisfaction with contact quantity week 6 | 3.76 (1.48) | 4.43 (1.48)
  Dissatisfaction with contact quantity week 7: number analyzed (Participants) | 29 | 34
  Dissatisfaction with contact quantity week 7 | 3.8 (1.44) | 4.36 (1.66)
  Dissatisfaction with contact quantity week 8: number analyzed (Participants) | 32 | 35
  Dissatisfaction with contact quantity week 8 | 3.74 (1.50) | 4.30 (1.54)
  Satisfaction with contact quantity Baseline (Average of Week 1 and 2) | 4.21 (1.34) | 4.3 (1.36)
  Satisfaction with contact quantity week 3: number analyzed (Participants) | 33 | 36
  Satisfaction with contact quantity week 3 | 4.13 (1.53) | 4.51 (1.55)
  Satisfaction with contact quantity week 4: number analyzed (Participants) | 30 | 36
  Satisfaction with contact quantity week 4 | 4.37 (1.32) | 4.31 (1.51)
  Satisfaction with contact quantity week 5: number analyzed (Participants) | 31 | 35
  Satisfaction with contact quantity week 5 | 4.3 (1.28) | 4.31 (1.48)
  Satisfaction with contact quantity week 6: number analyzed (Participants) | 32 | 35
  Satisfaction with contact quantity week 6 | 4.3 (1.36) | 4.36 (1.48)
  Satisfaction with contact quantity week 7: number analyzed (Participants) | 29 | 34
  Satisfaction with contact quantity week 7 | 4.09 (1.51) | 4.4 (1.37)
  Satisfaction with contact quantity week 8: number analyzed (Participants) | 32 | 35
  Satisfaction with contact quantity week 8 | 4.3 (1.55) | 4.2 (1.55)
  shared understanding Baseline (Average of Week 1 and 2) | 4.91 (1.38) | 4.77 (1.39)
  shared understanding week 3: number analyzed (Participants) | 33 | 36
  shared understanding week 3 | 4.72 (1.57) | 4.84 (1.46)
  shared understanding week 4: number analyzed (Participants) | 30 | 36
  shared understanding week 4 | 4.89 (1.21) | 4.75 (1.54)
  shared understanding week 5: number analyzed (Participants) | 31 | 35
  shared understanding week 5 | 4.96 (1.28) | 4.74 (1.59)
  shared understanding week 6: number analyzed (Participants) | 32 | 35
  shared understanding week 6 | 4.83 (1.36) | 4.79 (1.49)
  shared understanding week 7: number analyzed (Participants) | 29 | 34
  shared understanding week 7 | 4.93 (1.24) | 4.88 (1.43)
  shared understanding week 8: number analyzed (Participants) | 32 | 35
  shared understanding week 8 | 5.04 (1.23) | 4.79 (1.41)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting satisfaction with contact quality; Test type: Superiority; p = .04, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 2: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting dissatisfaction with contact quantity; Test type: Superiority; p = .44, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 3: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting satisfaction with contact quantity; Test type: Superiority; p = .99, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 4: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting knowing others' experience; Test type: Superiority; p = .87, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 5: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting shared understanding; Test type: Superiority; p = .98, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 6: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting relationship salience; Test type: Superiority; p = .76, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

4. Primary Outcome: UCLA Loneliness Scale
Description: The UCLA Loneliness Scale captures one's subjective feelings of loneliness over the past week for weekly surveys and over the past month for pretest and posttest surveys (20 items with ratings from 1 "Never" to 4 "Often"). The scores were averaged across the 20 items, with a score ranging from 1-4. A higher score indicates more loneliness.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Pretest | 2.21 (0.63) | 2.21 (0.73)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 2.08 (0.75) | 2.24 (0.76)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .29, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

5. Primary Outcome: Positive and Negative Affect Schedule (PANAS) (20 Items)
Description: Positive and Negative Affect Schedule (PANAS) (20 items) asks participants to report how often participants felt positive and negative feelings over the past week for weekly surveys, and over the past month for pre-test and post-test surveys. Scores were averaged across the items (Total positive and negative affect scores can range from 0-4, with a higher score indicating a higher level of positive affect or negative affect).
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Positive Affect Pretest | 2.32 (0.85) | 2.13 (0.93)
  Positive Affect Posttest: number analyzed (Participants) | 31 | 35
  Positive Affect Posttest | 2.14 (1.05) | 2.02 (1.03)
  Negative Affect Pretest | 1.09 (0.80) | 0.9 (0.67)
  Negative Affect Posttest: number analyzed (Participants) | 31 | 35
  Negative Affect Posttest | 1.00 (0.92) | 0.9 (0.74)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition predicting positive affect; Test type: Superiority; p = .51, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 2: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition predicting negative affect; Test type: Superiority; p = .83, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

6. Primary Outcome: Perceived Stress Scale (PSS)
Description: Perceived Stress Scale (PSS) asks participants' stress perception over the last month and scores were summed across the items (Possible scores range from 0 to 40 with higher scores indicating higher stress).
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Pretest | 23.08 (7.92) | 22.82 (8.66)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 22.32 (8.44) | 22.20 (7.78)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .51, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

7. Primary Outcome: Brief Symptom Inventory (BSI)
Description: Brief Symptom Inventory (BSI) captures participants' psychological distress over the past week, scores were summed across the items (Total score ranges from 0-72, with higher scores indicating more stress) (Derogatis, 1975).
Time Frame: Baseline (Average of Week 1 and 2), Weekly during the intervention from Week 3 to 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 35 | 36
units on a scale
  Baseline (Average of Week 1 and 2) | 19.26 (12.07) | 21.01 (12.67)
  Week 3: number analyzed (Participants) | 33 | 36
  Week 3 | 20.55 (13.09) | 20.17 (13.96)
  Week 4: number analyzed (Participants) | 30 | 36
  Week 4 | 20.4 (14.7) | 20.44 (13.76)
  Week 5: number analyzed (Participants) | 31 | 35
  Week 5 | 19.65 (14.88) | 19.8 (13.21)
  Week 6: number analyzed (Participants) | 32 | 35
  Week 6 | 18.72 (15.03) | 19.2 (13.75)
  Week 7: number analyzed (Participants) | 29 | 34
  Week 7 | 20.17 (16.08) | 19.32 (13.79)
  Week 8: number analyzed (Participants) | 31 | 35
  Week 8 | 17.71 (15.83) | 19.69 (14.03)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .65, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

8. Primary Outcome: Caregiver's Stress Scale
Description: Caregiver's Stress Scale has a series of subscales based on a conceptual model of caregivers' stress: overload, relational deprivation, job and caregiving conflict, role captivity, sense of self, caregiving competence, personal gain, management of situation, management of meaning, management of distress, and expressive support. Each subscale ranges from 1 (strongly disagree) to 4 (strongly agree), and each subscale was averaged (with possible score ranging from 1-4) so that higher scores would indicate a higher value.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Overload Pretest | 1.84 (0.92) | 1.61 (0.68)
  Overload Posttest: number analyzed (Participants) | 31 | 35
  Overload Posttest | 1.77 (0.80) | 1.58 (0.73)
  Relational Deprivation Pretest | 1.97 (0.97) | 1.83 (0.85)
  Relational Deprivation Posttest: number analyzed (Participants) | 31 | 35
  Relational Deprivation Posttest | 1.83 (0.86) | 1.83 (0.77)
  Job Caregiving Conflict Pretest | 2.18 (0.72) | 2.11 (0.60)
  Job Caregiving Conflict Posttest: number analyzed (Participants) | 31 | 35
  Job Caregiving Conflict Posttest | 2.25 (0.73) | 2.27 (0.75)
  Role Captivity Pretest | 1.88 (0.90) | 1.93 (0.83)
  Role Captivity Posttest: number analyzed (Participants) | 31 | 35
  Role Captivity Posttest | 1.82 (1.02) | 2.13 (1.04)
  Sense of Self Pretest | 3.66 (0.51) | 3.34 (0.58)
  Sense of Self Posttest: number analyzed (Participants) | 31 | 35
  Sense of Self Posttest | 3.55 (0.68) | 3.39 (0.57)
  Caregiving Competence Pretest | 3.34 (0.51) | 3.13 (0.75)
  Caregiving Competence Posttest: number analyzed (Participants) | 31 | 35
  Caregiving Competence Posttest | 3.32 (0.64) | 3.07 (0.60)
  Management of Situation Pretest | 2.84 (0.60) | 2.65 (0.63)
  Management of Situation Posttest: number analyzed (Participants) | 31 | 35
  Management of Situation Posttest | 2.73 (0.72) | 2.66 (0.47)
  Expressive Support Pretest | 3.16 (0.50) | 3.10 (0.41)
  Expressive Support Posttest: number analyzed (Participants) | 31 | 35
  Expressive Support Posttest | 3.12 (0.52) | 3.04 (0.61)
  Management of Distress Pretest | 2.18 (0.37) | 2.25 (0.35)
  Management of Distress Posttest: number analyzed (Participants) | 31 | 35
  Management of Distress Posttest | 2.37 (0.31) | 2.23 (0.39)
  Management of Meaning Pretest | 3.20 (0.52) | 2.94 (0.51)
  Management of Meaning Posttest: number analyzed (Participants) | 31 | 35
  Management of Meaning Posttest | 3.25 (0.44) | 2.97 (0.46)
  Personal Gain Pretest | 3.32 (0.65) | 2.93 (0.81)
  Personal Gain Posttest: number analyzed (Participants) | 31 | 35
  Personal Gain Posttest | 3.37 (0.70) | 2.98 (0.76)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting management of distress; Test type: Superiority; p = .01, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 2: Comparison: Social Exergame Treatment Group vs Control Group; time x condition interaction predicting caregiver overload; Test type: Superiority; p = .75, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 3: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting relational deprivation; Test type: Superiority; p = .59, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 4: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting job caregiving conflict; Test type: Superiority; p = .51, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 5: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting role captivity; Test type: Superiority; p = .25, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 6: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting sense of self; Test type: Superiority; p = .34, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 7: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting personal gain; Test type: Superiority; p = .75, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 8: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting caregiving competence; Test type: Superiority; p = .99, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 9: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting management of situition; Test type: Superiority; p = .61, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 10: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting management of meaning; Test type: Superiority; p = .92, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health
Statistical Analysis 11: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction predicting expressive support; Test type: Superiority; p = .96, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

9. Primary Outcome: International Physical Activity Questionnaire (IPAQ) Short Version
Description: International Physical Activity Questionnaire - Short Version. A continuous score was calculated expressed as MET (Metabolic Equivalents) minutes per week: Total MET-min/week = (Walk METs*min*days) + (Mod METs*min*days) + Vig METs*min*days). A higher score means a higher level of physical activity.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: Total METs minutes per week
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
Total METs minutes per week
  Pretest | 1523.69 (1324.89) | 1234.46 (1382.82)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 2066.86 (1482.13) | 1375.50 (1640.83)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .37, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

10. Secondary Outcome: Exercise Self-Efficacy
Description: 9 items assessed how certain participants will exercise under certain circumstances (e.g., when you are feeling under pressure or when you are away from home). Items are assessed from 1 (very sure) to 4 (not at all sure). Items were reverse coded and summed across all items with a score ranging from 9 to 36. A higher score indicates higher exercise self-efficacy.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Pretest | 19.74 (6.31) | 19.10 (6.99)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 22.87 (6.70) | 22.86 (6.68)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .89, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

11. Secondary Outcome: Satisfaction With Life Scale
Description: Items are assessed from 1 (disagree strongly) to 7 (agree strongly) summed across all items, ranging from 5-35. A higher score indicates a higher satisfaction with life.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Pretest | 19.84 (7.50) | 19.95 (7.95)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 20.61 (7.43) | 18.66 (8.73)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .30, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

12. Secondary Outcome: Sense of Control
Description: items were used to assess sense of control. For example: "There is little I can do to change many of the important things in my life." Items are assessed from 1 (strongly disagree) to 7 (strongly agree) and reverse coded. A sum across all items was calculated ranging from 6-42. A higher score indicates a higher sense of control.
Time Frame: Pretest (before week 1) and posttest (after week 8)
Population: N=38 in each condition completed the pretest. N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 38 | 38
score on a scale
  Pretest | 31.96 (6.05) | 29.77 (6.76)
  Posttest: number analyzed (Participants) | 31 | 35
  Posttest | 31.10 (7.32) | 29.07 (7.82)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Time x condition interaction; Test type: Superiority; p = .52, Mixed Models Analysis — Controlled for age, sex, education, and self-reported functional health

13. Secondary Outcome: Exergame Enjoyment Questionnaire (EEQ)
Description: Exergame Enjoyment Questionnaire (EEQ) was included in the posttest, which measured how much participants enjoyed the exergame (Fitzgerald et al., 2020). 20 items ranged from strongly disagree (1) to strongly agree (5) were summed. Scores rannged from 20 - 100, with a higher score indicating more exergame enjoyment.
Time Frame: Posttest (after week 8)
Population: N=31 in the treatment and N=35 in the control completed the posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Exergame Treatment Group | Control Group
Number analyzed (Participants) | 31 | 35
score on a scale | 67.29 (10.96) | 62.91 (13.67)
Statistical Analysis 1: Comparison: Social Exergame Treatment Group vs Control Group; Independent sample T-test comparing the treatment and control group; Test type: Superiority; p = .45, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 months
Description: any adverse event was documented and reported.
Arm/Group | Social Exergame Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 1/38 | 0/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Social Exergame Treatment Group (N=38) | Control Group (N=42)
Broken Ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 — the foot injury occurred at her workplace and does not appear to be related to her participation in the Study. The study involves walking and recording steps on a FitBit. The participant is no longer in the study as her mobility is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05032872/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT05032872/ICF_001.pdf